CLINICAL TRIAL: NCT05657795
Title: Does Closed-loop Automated Oxygen Control During Mechanical Ventilation Reduce the Duration of Supplementary Oxygen Treatment and the Amount of Time Spent in Hyperoxia? a Randomised Trial in Ventilated Infants Born At or Near Term
Brief Title: Optimising Neonatal Ventilation with Closed-loop Oxygen Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCH22-163
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Infant, Newborn, Diseases; Mechanical Ventilation Complication
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: Participating infants will be randomised either to manual oxygen control or closed-loop automated oxygen control, adjusted by clinical staff as necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual oxygen control (No Intervention): Standard ventilation with inspired oxygen concentration adjusted manually as per unit's protocol.
- Closed-loop automated oxygen control (Oxygenie, SLE 6000) (Other): Ventilation with Oxygenie software (closed-loop automated oxygen control system), adjusted by clinical staff as necessary
  Interventions: Device: Closed-loop automated oxygen control (Oxygenie, SLE6000)

INTERVENTIONS:
Device: Closed-loop automated oxygen control (Oxygenie, SLE6000) — The OxyGenie closed-loop oxygen saturation monitoring software (SLE) uses oxygen saturations from the SpO2 probe attached to the neonate, fed into an algorithm, to automatically adjust the percentage of inspired oxygen to maintain oxygen saturations within the target range. Manual adjustments including the percentage of FiO2 will be allowed at any point during the study if deemed appropriate by the clinical team.
  Arms: Closed-loop automated oxygen control (Oxygenie, SLE 6000)

SUMMARY:
Ventilated newborns frequently need supplemental oxygen but its use must be monitored carefully as both giving too much or too little oxygen can have harmful effects. Giving too little oxygen results to low oxygen levels (hypoxia) and increases the risk of complications and mortality. Excessive oxygen delivery (hyperoxia) increases the risk of diseases involving several organs such as the retinas and the lungs. Although infants born very preterm require support with their breathing more often, more mature neonates may also need to be ventilated at birth and to receive supplemental oxygen. Therefore, they may suffer from problems related to hypoxia and hyperoxia.

For the above reasons, oxygen levels are continuously monitored and the amount of oxygen provided is manually adjusted by the nurses and doctors.

Closed-loop automated oxygen control systems (CLAC) are a more recent approach that involves the use of a computer software added to the ventilator. This software allows for automatic adjustment of the amount of oxygen provided to the baby in order to maintain oxygen levels within a desired target range depending on the baby's age and clinical condition. Previous studies in preterm and very small infants showed that automated oxygen control systems provided the right amount of oxygen for most of the time and prevented hypoxia and hyperoxia with fewer manual adjustments required by clinical staff. Preliminary results from a study that included infants born at 34 weeks gestation and beyond showed that CLAC systems allowed to reduce the amount of supplementary oxygen more rapidly. With this study we aim to compare the time spent in hyperoxia and the overall duration of oxygen treatment between infants whose oxygen is adjusted either manually or automatically while they remain ventilated. This will help us understand if CLAC systems help reduce the complications related to oxygen treatment.

DETAILED DESCRIPTION:
This will be a randomised controlled trial. The investigators aim to recruit a minimum of forty ventilated infants born at or above 34 weeks of gestation. Participants will be randomised to either closed-loop automated oxygen control or manually controlled oxygen from recruitment to successful extubation.

Informed written consent will be requested from the parents or legal guardians of the infants and the attending neonatal consultant will be requested to assent to the study.

Eligible infants whose parents consent to the study will be enrolled within 24 hours of initiation of mechanical ventilation.

Randomisation will be performed using an online randomisation generator. Patients will be ventilated using SLE6000 ventilators. Ventilator settings will be manually adjusted by the clinical team as per unit's protocol. The intervention group, in addition to standard care will also be connected to the Oxygenie closed-loop oxygen saturation monitoring software (SLE). This software uses oxygen saturations from the SpO2 probe attached to the neonate, fed into an algorithm, to automatically adjust the percentage of inspired oxygen to maintain oxygen saturations within the target range. Manual adjustments to the inspired oxygen concentration will be allowed at any point during the study if deemed appropriate by the clinical team.

Patient will be studied from enrolment till successful extubation. If an infant fails extubation and required reintubation within 48 hours, he will be studied in his initial study arm. Therefore, for the infants randomised at the intervention group CLAC will resume.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at or above 34 weeks completed gestation requiring mechanical ventilation and admitted to King's NICU within 24 hours of initiation of mechanical ventilation.

Exclusion Criteria:

* Preterm infants less than 34 weeks gestation
* Infants with cyanotic congenital heart disease
* Infants on high frequency oscillatory ventilation (HFOV)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The duration of oxygen treatment | Through study completion, an average of 1 year
  The duration of oxygen treatment will be measured in median (interquartile range) number of days of oxygen treatment for participants in each group.
The percentage of time spent in hyperoxia | Through study completion, an average of 1 year
  Target oxygen saturation range for our study population is 92-96%. Hyperoxia is defined as the time spent with oxygen saturation levels exceeding 96%. The time spent in hyperoxia will be calculated as a percentage of the total time of monitoring.

SECONDARY OUTCOMES:
The percentage of time spent receiving an inspired oxygen concentration (FiO2) above 30% | Through study completion, an average of 1 year
  The time spent with an FiO2>30% will be calculated as a percentage of the total time of monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Dassios, PhD, Principal Investigator — King's College Hospital/ King's College London
Locations (1):
- King's College Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramadan G, Paul N, Morton M, Peacock JL, Greenough A. Outcome of ventilated infants born at term without major congenital abnormalities. Eur J Pediatr. 2012 Feb;171(2):331-6. doi: 10.1007/s00431-011-1549-8. Epub 2011 Aug 11. PMID 21833494
- [Background] Williams LZJ, McNamara D, Alsweiler JM. Intermittent Hypoxemia in Infants Born Late Preterm: A Prospective Cohort Observational Study. J Pediatr. 2019 Jan;204:89-95.e1. doi: 10.1016/j.jpeds.2018.08.048. Epub 2018 Oct 1. PMID 30287066
- [Background] Lakshminrusimha S, Konduri GG, Steinhorn RH. Considerations in the management of hypoxemic respiratory failure and persistent pulmonary hypertension in term and late preterm neonates. J Perinatol. 2016 Jun;36 Suppl 2:S12-9. doi: 10.1038/jp.2016.44. PMID 27225960
- [Background] Salverda HH, Cramer SJE, Witlox RSGM, Dargaville PA, Te Pas AB. Automated oxygen control in preterm infants, how does it work and what to expect: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2021 Mar;106(2):215-221. doi: 10.1136/archdischild-2020-318918. Epub 2020 Jul 30. PMID 32732378
- [Background] Sturrock S, Ambulkar H, Williams EE, Sweeney S, Bednarczuk NF, Dassios T, Greenough A. A randomised crossover trial of closed loop automated oxygen control in preterm, ventilated infants. Acta Paediatr. 2021 Mar;110(3):833-837. doi: 10.1111/apa.15585. Epub 2020 Oct 6. PMID 32969040
- [Background] Abdo M, Hanbal A, Asla MM, Ishqair A, Alfar M, Elnaiem W, Ragab KM, Nourelden AZ, Zaazouee MS. Automated versus manual oxygen control in preterm infants receiving respiratory support: a systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6069-6076. doi: 10.1080/14767058.2021.1904875. Epub 2021 Apr 8. PMID 33832390
- [Derived] Kaltsogianni O, Dassios T, Jenkinson A, Greenough A. Does closed-loop automated oxygen control reduce the duration of supplementary oxygen treatment and the amount of time spent in hyperoxia? A randomised controlled trial in ventilated infants born at or near term. Trials. 2023 Jun 15;24(1):404. doi: 10.1186/s13063-023-07415-9. PMID 37316885